CLINICAL TRIAL: NCT00374985
Title: Prospective, Open, Multicentre Phase I/II Study to Evaluate the Safety and Efficacy of a Neoadjuvant Radiochemotherapy With Docetaxel and Oxalipaltin in Patients With Adenocarcinoma of the Gastric-oesophageal Junction
Brief Title: Safety and Efficacy of Neoadjuvant Radiochemotherapy in Adenocarcinoma of the Gastric-oesophageal Junction
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, PD Dr Markus Möhler, Professor, Johannes Gutenberg University Mainz
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC-DOR-2004
Record Dates: First submitted 2006-09-11; First posted 2006-09-12 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Esophageal Neoplasms; Stomach Neoplasms
Keywords: chemoradiation; docetaxel; oxaliplatin; gastric; neoadjuvant; radiochemotherapy
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — Docetaxel; Oxaliplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- one arm (Experimental)
  Interventions: Drug: Docetaxel, Oxaliplatin; Procedure: Radiotherapy

INTERVENTIONS:
Drug: Docetaxel, Oxaliplatin — weekly doses
Procedure: Radiotherapy — regular fractions

SUMMARY:
The purpose of this study is to determine the dose limiting toxicity and the maximum tolerable dose of the radiochemotherapy with Docetaxel and Oxaliplatin in patients with adenocarcinoma of the gastric-oesophageal junction.

DETAILED DESCRIPTION:
Radiotherapy starts on day 1 of chemotherapy after the application of Docetaxel and Oxaliplatin and will be administered in single doses of 1.8 Gy once daily and five times a week for 5 weeks.

In the sixth treatment week a boost of 3 further radiations with 1.8 Gy will be applied.

Simultaneous chemotherapy:

Initially, in part A of the study the maximum tolerable dose (MTD) for the simultaneous chemotherapy will be identified with a 3-step dose escalation scheme:

Level 1: Docetaxel: 20 mg/m2 Oxaliplatin 40 mg/m2 i.v., Level 2: Docetaxel: 20 mg/m2 Oxaliplatin 50 mg/m2 i.v., Level 3: Docetaxel: 25 mg/m2 Oxaliplatin 50 mg/m2 i.v.,

The treatment starts with 3 patients in level 1. If no dose limiting toxicities appear, it will be switched to dose level 2. The same applies for the switch from level 2 to level 3. If a DLT appears on one level, a further 3 patients will be treated within this dose level.

If in one level at least 2 of 6 patients show DLT, the subjacent level will be defined as the maximum tolerable dose (MTD).

ELIGIBILITY:
Inclusion Criteria:

* adenocarcinoma of gastric-esophagal junction
* stage II to III
* unidimensional measurable disease

Exclusion Criteria:

* surgery of primary tumor
* metastasis
* prior chemo- or radiotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
maximum tolerable dose and safety | until August 2010

CONTACTS AND LOCATIONS:
Overall Officials: Markus Moehler, MD, Principal Investigator — Johannes Gutenberg University Mainz
Locations (1):
- Johannes-Gutenberg-Universität, Mainz, Rhineland-Palatinate, Germany

REFERENCES:
- [Derived] Moehler M, Gockel I, Roessler HP, Arnold D, Trarbach T, Thomaidis T, Klautke G, Rodel C, Brenner B, Lang H, Galle PR, Schimanski CC, Schmidberger H. Prospective, open, multi-centre phase I/II trial to assess safety and efficacy of neoadjuvant radiochemotherapy with docetaxel and oxaliplatin in patients with adenocarcinoma of the oesophagogastric junction. BMC Cancer. 2013 Feb 11;13:75. doi: 10.1186/1471-2407-13-75. PMID 23394629